CLINICAL TRIAL: NCT00984529
Title: Evaluation of Clinical Signs and Symptoms of Chronic Heart Failure in Patients Treated With Candesartan Cilexetil in Croatia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MCMD, AstraZeneca
Other Study IDs: NIS-CHR-ATA-2008/1
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Heart Failure
Keywords: Chronic heart failure; candesartan cilexetil; clinical signs; symptoms
MeSH Terms: conditions — Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Cardiologist´s office patients

SUMMARY:
The purpose of this study is to determine whether treatment with candesartan cilexetil for at least 6 months in patients with chronic heart failure improves clinical signs and symptoms of chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed chronic heart failure
* Patients treated for at least 6 months with candesartan cilexetil
* Signed Informed consent

Exclusion Criteria:

* Hypersensitivity to candesartan cilexetil
* Pregnancy / lactation
* Severe hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate clinical signs and symptoms of chronic heart failure (in terms of NYHA status, fluid retention and tiredness/fatigue) after at least 6 months of treatment with candesartan cilexetil | 1 visit (after at least 6 months of treatment)

SECONDARY OUTCOMES:
To evaluate ventricular function after at least 6 months of treatment with candesartan cilexetil | 1 visit (after at least 6 months of treatment)
To gain insight into usage of candesartan cilexetil in real life for chronic heart failure in Croatia | 1 visit (after at least 6 months of treatment)
To evaluate patient's compliance with prescribed treatment | 1 visit (after at least 6 months of treatment)

CONTACTS AND LOCATIONS:
Locations (15):
- Croatia (15):
  - Research Site, Biograd na Moru
  - Research Site, Bjelovar
  - Reserach Site, Čakovec
  - Research Site, Karlovac
  - Reserach Site, Krapinske Toplice
  - Research Site, Novi Marof
  - Research Site, Opatija
  - Research Site, Osijek
  - Research Site, Pula
  - Research Site, Rijeka
  - Reserach Site, Sl. Brod
  - Research Site, Split
  - Research Site, Stubičke Toplice
  - Reserach Site, Zabok
  - Research Site, Zagreb